CLINICAL TRIAL: NCT03059628
Title: Evaluation of a Personalized Normative Feedback Repeatedly Delivered Via a Mobile Application After a Brief Therapeutic Intervention on Alcohol-related Risks: a Multi Center Randomized Open Study in Young Adults Admitted to Emergency Room for Acute Alcohol Intoxication (AAI).
Brief Title: Evaluation of a Personalized Normative Feedback Repeatedly Delivered Via a Mobile Application After a Brief Therapeutic Intervention on Alcohol-related Risks:
Acronym: IFACAP
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The number of participants included and especially who connected to the application (less than 50% of the target) does not meet the objective set by the study.
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 35RC15_8976_IFACAP
Record Dates: First submitted 2017-02-16; First posted 2017-02-23 (Actual); Last update posted 2019-03-27 (Actual); Status verified 2019-03

CONDITIONS: Acute Alcohol Intoxication
MeSH Terms: conditions — Alcoholic Intoxication | interventions — Patient Health Questionnaire

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Personalized Normative Feedback group (Experimental): A personalized normative feedback using a tablet application will be performed after the BTI at ED. The application installed on the patient's smartphone will automatically repeat the PNF, using a local algorithm, once a month over a 6-months period after discharge, and once every two months in the following 6-month period. It will be also possible to perform the PNF on the server website.
  Interventions: Other: Personalized Normative Feedback; Other: Brief Therapeutic Intervention; Other: Evaluation questionnaire
- Control group (Other): The control group will not receive further counseling or information after the baseline BTI at ED. The application installed in this group will be only used for the evaluation questionnaire at 6 and 12 months
  Interventions: Other: Brief Therapeutic Intervention; Other: Evaluation questionnaire

INTERVENTIONS:
Other: Personalized Normative Feedback — This "PNF" technique use information designed to correct normative misperceptions to reduce heavy drinking. Much of the alcohol consumption among college students stems from the fairly widespread perception that one's peers expect regular and sometimes extreme drinking participation (subjective drinking norms). The PNF approach is designed to counter this perception by giving students accurate figures on how much their peers actually drink (actual drinking norms). It also aims to improve students' understanding of alcohol use in general and the firmly established negative outcomes associated with short - and long-term patterns of excessive drinking.
  Arms: Personalized Normative Feedback group
Other: Brief Therapeutic Intervention — BTI are brief (typically one session 20-30 mns) and incorporate some or all of the following elements:feedback on the person's alcohol use and any alcohol-related harm; clarification as to what constitutes low risk alcohol consumption; information on the harms associated with risky alcohol use; benefits of reducing intake; motivational enhancement; analysis of high risk situations for drinking and coping strategies; and the development of a personal plan to reduce consumption.
Other: Evaluation questionnaire — The patient have to fill the same evaluation questionnaire at J0, M6 and M12

SUMMARY:
BTI (Brief Therapeutic Intervention) motivates individuals admitted to ED (Emergency Department) for acute intoxication to take actions to prevent further alcohol-related issues. The present project aims at underpinning this intervention by actively involving patients in the monitoring of their alcohol-related risk following discharge. While several web-based preventive interventions towards alcohol already exist, the repeated delivering of PNF (Personalized Normative Feedback) using mobile technology after a BTI constitutes a novel approach to reduce alcohol-related harms. Investigators propose to test the effect of a mobile PNF following a BTI delivered by a psychologist during an ED visit for alcohol intoxication. The mobile PNF will be additionally delivered once a month in the 6-months period after discharge, and once every two months in the following 6-month period, via a smartphone application connected to a central server. The study will include 18-26 years old adults, as this population includes most active students and is often lost to follow-up after ED visits; and aims the reduction of heavy drinking occasions, as this issue account for most of alcohol-related ED visits in this population.

DETAILED DESCRIPTION:
The study will begin simultaneously in all the centers, in September, at the beginning of the university year. When patients will be admitted in the ED for alcohol intoxication, they will first meet the entry nurse, who will make the orientation as usual. Participants will be marked as eligible for the study, and a breath test or a blood alcohol test will be performed. On the following morning, a psychologist will evaluate all potential patients, and check the inclusion criteria. In case of eligibility, the study procedure will be explained and the patient and a medical doctor present in the ED will sign an informed consent. The patient will be included and a baseline assessment will be performed using a web-based questionnaire implemented on a digital tablet. These inputs will automatically generate an identification number and a personal dashboard on a centralized server. Individual codes will be also given to each patient for accessing their personal dashboard on the server from a home computer. The patient will then be randomized, with stratification on center, sex, and absence or presence of a daily consumption of cannabis, between the intervention and the control groups. The psychologist will then perform a brief therapeutic intervention for both groups. Investigators plan to train all psychologists all together to the brief intervention. Then a smartphone application will be installed on the patient's smartphone. Follow-up assessments will be conducted 6 and 12 months after baseline using the same questionnaire, through the smartphone application or on the server website. The application will recall the patient by the means of automatic notifications at 6 and 12 months. Data will be push to the server with the identification number, without any other nominal information. In case patients do not perform the evaluation one week after the expected date, they will be contacted by any means (telephone, postal mail, email or SMS with a link to the software) by a research assistant to recall them to do the evaluation. Participants will be compensated using gift vouchers for the time lost for the interview.

Experimental group :

A personalized normative feedback using a tablet application will be performed after the BTI at ED. The application installed on the patient's smartphone will automatically repeat the PNF, using a local algorithm, once a month over a 6-months period after discharge, and once every two months in the following 6-month period. It will be also possible to perform the PNF on the server website.

Control group :

Patients in the control group will receive the BTI at the ED. The application installed on this group will only realize the evaluation questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-26 years;
* Admitted for an acute alcohol intoxication to the ED from Thursday to Sunday;
* Need to be kept in the ED for detoxification;
* Alcohol breath test or blood alcohol concentration if breath test impossible greater than 0.5 gram per liter at the admission to the ED;
* Able to understand and remember the component of the study;
* Use of a smartphone;
* Written informed consent.

Exclusion Criteria:

* Patients in police custody and not admitted to emergency;
* Patients admitted for suicidal ideation or attempt;
* Injury requiring an hospitalization;
* Additional need for psychiatric or addiction evaluation;
* Current care in addiction facilities (last contact less than 3 months);
* Planning of a specialized care at the end of the hospitalization;
* Persons participant to major legal protection (safeguarding justice, guardianship, trusteeship), persons deprived of liberty.
* Patients participating in another interventional research

Ages: 18 Years to 26 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 222 (Actual)
Dates: Start 2017-09-22 (Actual); Primary Completion 2018-10-28 (Actual); Study Completion 2018-10-28 (Actual)

PRIMARY OUTCOMES:
Reduction of the number of heavy drinking occasions | at 12 months
  Reduction (expressed as a percentage) of the number of heavy drinking occasions (= 7 or more standard drinks of 10 g pure alcohol in one occasion) in the precedent month between baseline (nbaseline) and the evaluation done 12 months after the admission in the ED (n12 months) :
  Change = (nbaseline - n12months) / nbaseline

SECONDARY OUTCOMES:
Reduction of the number of standard drinks | at 6 months and at 12 months
  Reduction of the number of standard drinks per heavy drinking occasions in the month before the evaluation (done 6 and 12months after the admission in the ED) versus the number at baseline (in the month before the admission to the ED);
Reduction of the number of heavy drinking occasions | at 6 months
  Reduction of the number of heavy drinking occasions in the month before the evaluation (done 6 months after the admission in the ED) versus the number at baseline (in the month before the admission to the ED);
Reduction of the number of alcohol intoxications | at 6 months and at 12 months
  Reduction of the number of alcohol intoxications (participantively defined by the patient as drunkenness) in the month before the evaluation (done 6 and 12 months after the admission in the ED) versus the number at baseline (in the month before the admission to the ED);
Reduction of the number of binge drinking | at 6 months and at 12 months
  Reduction of the number of binge drinking (see definition above) in the month before the evaluation (done 6 and 12 months after the admission in the ED) versus the number at baseline (in the month before the admission to the ED);
Reduction of total alcohol consumption | at 6 months and at 12 months
  Reduction of total alcohol consumption (in mean standard drinks per week) in the month before the evaluation (done 6 and 12 months after the admission in the ED) versus the number at baseline (in the month before the admission to the ED);
Alcohol related problems | at 6 months and at 12 months
  Alcohol related problems in the 6 months and in the year before the evaluations
Hospitalisations or admissions in the ED, injuries, violence, unwanted or unprotect sexual behaviours, loss of employment or school problems. | at 6 months and at 12 months
  Hospitalisations or admissions in the ED, injuries, violence, unwanted or unprotect sexual behaviours, loss of employment or school problems.

CONTACTS AND LOCATIONS:
Overall Officials: Romain MOIRAND, MD/PHD, Principal Investigator — Rennes Pontchaillou Hospital
Locations (5):
- France (5):
  - Centre Hospitalier Universitaire Amiens Picardie, Amiens
  - Centre Hospitalier Universitaire Angers, Angers
  - Hôpital Saint André, Bordeaux
  - Centre Hospitalier Universitaire Rennes Pontchaillou, Rennes
  - Centre Hospitalier Régional Universitaire de Tours - Hôpital trousseau, Tours